CLINICAL TRIAL: NCT04615117
Title: An Outcomes Study Utilizing Allomend(R) HD for Superior Capsular Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Orthopaedics Research and Education Foundation (Other)
Collaborators: AlloSource (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLOMEND
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tear or Rupture, Not Specified as Traumatic
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients treated with Superior Capsular Reconstruction with Allomend

SUMMARY:
Rotator cuff tears can usually be repaired with excellent results, however some chronic, extensive rotator cuff tears are not reparable secondary to tendon retraction with inelasticity, muscle atrophy, and fatty infiltration. Arthroscopic superior capsular reconstruction (SCR) utilizing allograft or autograft tissue has been shown to restore superior glenohumeral stability and function of the shoulder joint in patients with irreparable rotator cuff tears. Grafts utilized for SCR have included fascia lata, hamstring autograft, human acellular dermal tissue matrix (HADTM), and acellular porcine dermal xenograft. Due to donor morbidity associated with autografts and the graft rejection potential of xenograft, HADTM has become a common graft of choice for SCR. The purpose of this study is to determine if patients treated with SCR using AlloMend have acceptable clinical and anatomic outcomes.

DETAILED DESCRIPTION:
Rotator cuff tears can usually be repaired with excellent results, however some chronic, extensive rotator cuff tears are not reparable secondary to tendon retraction with inelasticity, muscle atrophy, and fatty infiltration. Arthroscopic superior capsular reconstruction (SCR) utilizing allograft or autograft tissue has been shown to restore superior glenohumeral stability and function of the shoulder joint in patients with irreparable rotator cuff tears.Grafts utilized for SCR have included fascia lata, hamstring autograft, human acellular dermal tissue matrix (HADTM), and acellular porcine dermal xenograft. Due to donor morbidity associated with autografts and the graft rejection potential of xenograft, HADTM has become a common graft of choice for SCR. The purpose of this study is to determine if patients treated with SCR using AlloMend have acceptable clinical and anatomic outcomes. We predict there will be significant improvement in radiographic, clinical, and patient reported outcomes in patients undergoing SCR for extensive, primarily irreparable rotator cuff tears when AlloMend allograft is utilized.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are undergoing SCR for massive rotator cuff
* Adult patients (≥18)
* Pre-operative MRI obtained within 26 weeks prior to surgery
* Must have 3 out of 5 external rotation strength
* Must have intact teres minor

Exclusion Criteria:

* Worker's Compensation Case
* Persons with a mental or cognitive disability deemed significant enough that they would not be capable of complying with a restricted rehabilitation program or completing the outcome measures
* Patients with known contraindications to MRI
* Pectoralis major, pectoralis minor, deltoid, or latissimus dorsi dysfunction
* Acute fractures of humerus, clavicle, scapula
* Inability to speak and/or understand English

Intra-Op Exclusion Criteria:

* Anterosuperior escape of the glenohumeral joint due to a completely incompetent anterosuperior cuff and coracoacromial ligament (CAL)
* Unable to fix the graft on the humeral side utilizing a double row repair
* Inability to address subscapularis pathology
* Diffuse bipolar cartilage loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with massive rotator cuff tears
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acromiohumeral interval change | 24 months
  Xrays will be used to compare the amount of superior humeral migration between 12 month xrays and 24 month xrays
Clinical Failure | Within 24 months
  Revision Surgery
Rotator Cuff Integrity and Graft Incorporation | 24 months
  These will be assessed via MRI with Arthrogram- changes will be compared between the 12 and 24 month time points

SECONDARY OUTCOMES:
Function (Activities of Daily Living) | 24 months
  Function will be assessed via the American Shoulder and Elbow Score (0-100; higher score is better)
Function (Overall Normal rating) | 24 months
  Function will be assessed via the Single Assesment Numeric Evaluation (SANE) (0-100; where 100 is normal)
Shoulder Pain | 24 months
  Pain will be assessed on a Visual Analog Scale (VAS) (0-10; where 0 is no pain and 10 is the worst pain imaginable)
Range of Motion | 24 months
  Function will be assessed by measuring active range of motion (forward flexion, abduction, external rotation, internal rotation) with a goniometer
Resilience | 24 months
  Resilience will be assessed via the Brief Resilience Score (BRS) (scores 1-5; higher score = higher resilience)

CONTACTS AND LOCATIONS:
Overall Officials: Armodios Hatzidakis, MD, Principal Investigator — Western Orthopaedics Education and Research Foundation
Locations (1):
- Western Orthopaedics Education and Research Foundation, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
aggregate data

REFERENCES:
- [Result] Mihata T, McGarry MH, Kahn T, Goldberg I, Neo M, Lee TQ. Biomechanical Role of Capsular Continuity in Superior Capsule Reconstruction for Irreparable Tears of the Supraspinatus Tendon. Am J Sports Med. 2016 Jun;44(6):1423-30. doi: 10.1177/0363546516631751. Epub 2016 Mar 4. PMID 26944572
- [Result] Adams CR, Denard PJ, Brady PC, Hartzler RU, Burkhart SS. The Arthroscopic Superior Capsular Reconstruction. Am J Orthop (Belle Mead NJ). 2016 Jul-Aug;45(5):320-4. PMID 27552457
- [Result] Pennington WT, Bartz BA, Pauli JM, Walker CE, Schmidt W. Arthroscopic Superior Capsular Reconstruction With Acellular Dermal Allograft for the Treatment of Massive Irreparable Rotator Cuff Tears: Short-Term Clinical Outcomes and the Radiographic Parameter of Superior Capsular Distance. Arthroscopy. 2018 Jun;34(6):1764-1773. doi: 10.1016/j.arthro.2018.01.009. Epub 2018 Feb 15. PMID 29456069
- [Result] Polacek M. Arthroscopic Superior Capsular Reconstruction With Acellular Porcine Dermal Xenograft for the Treatment of Massive Irreparable Rotator Cuff Tears. Arthrosc Sports Med Rehabil. 2019 Nov 13;1(1):e75-e84. doi: 10.1016/j.asmr.2019.08.001. eCollection 2019 Nov. PMID 32266343
- [Result] Burkhart SS, Pranckun JJ, Hartzler RU. Superior Capsular Reconstruction for the Operatively Irreparable Rotator Cuff Tear: Clinical Outcomes Are Maintained 2 Years After Surgery. Arthroscopy. 2020 Feb;36(2):373-380. doi: 10.1016/j.arthro.2019.08.035. Epub 2019 Dec 18. PMID 31864817